CLINICAL TRIAL: NCT07182721
Title: A Phase II, Single-Arm, Single-Center, Prospective Study of SKB264 Plus Inetetamab in HER2-Positive Unresectable Locally Advanced or Metastatic Breast Cancer Patients Progressing After T-DXd Treatment
Brief Title: SKB264 Plus Inetetamab in HER2-Positive Metastatic Breast Cancer Patients Progressing After T-DXd Treatment
Acronym: SHINE-HER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Hongxia Wang, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2505320-11-2507
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive, Unresectable, Locally Advanced or Metastatic Breast Cancer; SKB264; Inetetamab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- metastatic HER2-positive breast cancer (Experimental): Patients with HER2-positive, unresectable, locally advanced or metastatic breast cancer previously treated with and refractory to T-DXd
  Interventions: Drug: SKB264 Plus Inetetamab

INTERVENTIONS:
Drug: SKB264 Plus Inetetamab — SKB264: 5 mg/kg administered on Day 1 of each 2-week cycle. Inetetamab: an initial loading dose of 6 mg/kg is administered, followed by subsequent maintenance doses of 4 mg/kg. Dosing occurs on Day 1 of each 2-week cycle.

SUMMARY:
This is a prospective, single-arm, single-center, Phase II clinical study designed to assess the preliminary efficacy and safety of SKB264 Plus Inetetamab plus inetetamab for the treatment of HER2-positive, unresectable, locally advanced or metastatic breast cancer following progression on prior T-DXd therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female.
2. Patients with histologically or cytologically confirmed breast cancer who meet the following criteria:

   1. Unresectable locally advanced or metastatic breast cancer.
   2. Pathologically confirmed HER2-positive breast cancer, regardless of hormone receptor (HR) status. HER2 positivity is defined as: IHC 3+, or IHC 2+ and FISH positive.
   3. Prior treatment for unresectable locally advanced or metastatic disease must have included the following anti-HER2 therapies: trastuzumab deruxtecan (T-DXd) and trastuzumab (or a trastuzumab biosimilar). Patients who received T-DXd and trastuzumab (or a biosimilar) in the (neo)adjuvant setting and experienced recurrence or metastasis during or within 12 months of completing therapy are eligible. Additionally, prior treatment regimens must have included a taxane.
   4. Documented disease progression or unacceptable toxicity after the last line of therapy for unresectable locally advanced or metastatic disease.
3. ECOG performance status of 0-2, with a life expectancy of > 3 months.
4. At least one measurable target lesion according to RECIST v1.1 criteria.
5. Adequate organ and bone marrow function, as defined below:

   1. Complete Blood Count: Absolute Neutrophil Count (ANC) ≥ 1.5 × 10⁹/L; Platelets ≥ 75 × 10⁹/L; Hemoglobin ≥ 90 g/L.
   2. Liver Function: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 3.0 × upper limit of normal (ULN); Total bilirubin (TBIL) ≤ 1.5 × ULN. For patients with liver metastases, ALT and AST ≤ 5.0 × ULN.
   3. Renal Function: Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (calculated by the Cockcroft-Gault formula).
   4. Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 × ULN and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.
   5. Echocardiogram: Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
   6. 12-lead ECG: QT interval corrected by Fridericia's formula (QTcF) < 470 ms for females and < 450 ms for males.
6. Voluntarily agrees to participate in the study by signing the informed consent form (ICF), and is willing and able to comply with follow-up procedures.

Exclusion Criteria:

1. Meningeal metastases confirmed by MRI or lumbar puncture.
2. Presence of spinal cord compression or clinically active central nervous system (CNS) metastases (defined as untreated or symptomatic metastases, or those requiring corticosteroids or anticonvulsants to control associated symptoms). Patients with previously treated brain metastases may be enrolled, provided they are clinically stable for at least 4 weeks, have no imaging evidence of progression, and at least 2 weeks have passed since the completion of brain radiotherapy and the discontinuation of corticosteroids or anticonvulsants for this indication.
3. Presence of third-space fluid accumulation (e.g., significant pleural effusion) that cannot be controlled by drainage or other methods.
4. Prior treatment with inetetamab or any TROP-2 antibody-drug conjugate (ADC).
5. Receipt of whole-brain radiotherapy, chemotherapy, biologic targeted therapy, immunotherapy, surgery, endocrine therapy, or other investigational drugs within 2 weeks prior to the first dose of study treatment.
6. Concurrent treatment with any other anti-cancer therapy.
7. Known history of hypersensitivity to any component of the study drugs. Permanent discontinuation of prior trastuzumab or its biosimilars due to any toxicity.
8. Severe or uncontrolled cardiac disease requiring treatment, including:

   1. Congestive heart failure of New York Heart Association (NYHA) Class 3 or 4.
   2. Unstable angina pectoris uncontrolled by medication.
   3. Myocardial infarction within 6 months prior to the first dose of study treatment.
   4. Severe arrhythmia requiring medical treatment (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
   5. History of symptomatic congestive heart failure or a Left Ventricular Ejection Fraction (LVEF) <40% during previous trastuzumab therapy.
9. Presence of any severe concomitant disease that, in the investigator's judgment, could jeopardize patient safety or interfere with study completion (e.g., uncontrolled severe diabetes, hypertension, autoimmune diseases), or any other condition deemed unsuitable for enrollment by the investigator.
10. Toxicity from prior anti-cancer therapy that has not resolved to NCI-CTCAE v5.0 Grade ≤1 or baseline level (with the exception of Grade 2 alopecia, pigmentation, or other toxicities such as simple laboratory abnormalities that the investigator considers to pose no safety risk).
11. History of other malignancies within the past 5 years, with the exception of curatively treated carcinoma in-situ, basal cell or squamous cell skin carcinoma, or papillary thyroid carcinoma after curative resection.
12. History of immunodeficiency, including a positive HIV test, active Hepatitis B or C, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
13. Known history of neurological or psychiatric disorders, including epilepsy or dementia.
14. Female patients of childbearing potential who are pregnant or breastfeeding. A negative serum pregnancy test is required within 7 days prior to randomization. Patients of childbearing potential must agree to use a highly effective method of contraception throughout the study and for 7 months after the last dose of study drug.
15. Any other condition that, in the opinion of the investigator, would make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator | At baseline, at the time point of every 6 weeks, up to 1 years
  ORR (Objective response rate) is the percentage of evaluable patients with a confirmed investigator-assessed response of CR (complete response) or PR (partial response) per RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No